CLINICAL TRIAL: NCT06669884
Title: Use of Determine Learning-based Cardiodynamicsgram (CDG) for Rapid and Precise Stratification of Chest Pain in Emergency Department
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: QLEmer-CDG-1
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Chest Pain; Acute Coronary Syndrome
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- machine learning algorithm: machine learning algorithm based on ECG features
  Interventions: Other: Cardiodynamicsgram (CDG)

INTERVENTIONS:
Other: Cardiodynamicsgram (CDG) — Cardiodynamicsgram (CDG) technique

SUMMARY:
Chest pain accounts for 10-20 percent of all emergency department visits. The stratification of chest pain is always a challenge. Electrocardiograms (ECG) have been used in clinical practice for 100 years, which is too important to be replaced due to its advantages of non-invasive, simple, rapid and inexpensive. ECG contains numerous signals derived from depolarization and repolarization of cardiomyocytes. However, the interpretation of ECG hasn't improved much in a hundred years. Based on determine-learning, Cong W's team developed an technique called "cardiodynamicsgram (CDG)", which is an outstanding method to identify myocardial ischemia. This study will further investigate the accuracy of CDG in stratification of patients with chest pain in Emergency department.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* Those with suspected ACS who have symptoms of acute chest pain, visiting in the emergency department

Exclusion Criteria:

* Those who diagnosed with ST-segment elevation myocardial infarction (STEMI)
* Those with hemodynamic instability (cardiogenic shock, cardiac arrest)
* Those with malignant arrhythmias(ventricular tachycardia, ventricular fibrillation, third-degree atrioventricular block)
* Those with aortic coarctation, or acute pulmonary embolism
* Those who has an unanalysable ECG report due to loosened leads, unstable baseline, or signal interference, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who suffers from acute chest pain suspected with acute coronary syndrome (ACS)
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of CDG in the risk stratification of patients who have symptoms of acute chest pain suspected with acute coronary syndrome （ACS) | from the date of enrollment until the date of discharge, up to 30 days
  Establishing an algorithm model of CDG in risk stratification in chest pain patients, the efficacy of the model was assessed by sensitivity, specificity, accuracy, positive predictive value, negative predictive value, and AUC, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China